CLINICAL TRIAL: NCT01333826
Title: Does Schooling Protect Young Women From HIV?
Brief Title: Schooling, Income, and HIV Risk in Malawi
Acronym: SIHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: World Bank (Other); University of California, San Diego (Other); University of Malawi (Other)
Responsible Party: Principal Investigator, Sarah Baird, Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KCP: RF-P109215-RESE-TF090932; RSB: RF-P109215-RESE-BBRSB (Other Grant/Funding Number: World Bank)
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: HIV; Schooling; Conditional Cash Transfers; Unconditional Cash Transfers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unconditional cash transfers (Experimental): Monthly cash transfers given to households with school aged girls with no strings attached. Transfer amounts randomized within this arm.
  Interventions: Behavioral: Zomba Cash Transfer Program
- Conditional Cash Transfer (Experimental): Monthly cash transfers given to households with school aged girls conditional on regular school attendance (80%). Transfer amounts randomized within this arm.
  Interventions: Behavioral: Zomba Cash Transfer Program
- Control Group (No Intervention): No cash transfer program implemented in this group.

INTERVENTIONS:
Behavioral: Zomba Cash Transfer Program — Cash transfers were provided monthly to a randomly selected sample of school aged girls. Amounts were also varied in both treatment arms.
  Arms: Conditional Cash Transfer; Unconditional cash transfers

SUMMARY:
This study is designed to evaluate a two-year randomized intervention in Malawi that provides cash transfers to current schoolgirls (and young women who have recently dropped out of school) to stay in (and return to) school in order to understand the possible effects of such programs on the sexual behavior of the beneficiaries and their subsequent HIV risk.

DETAILED DESCRIPTION:
Motivation:

Education has been suggested as a "social vaccine" to prevent the spread of HIV (Jukes, Simmons, and Bundy, 2008), but almost all of the evidence we have on the link between school attendance (or attainment) and the risk of HIV infection comes from cross-sectional studies. Furthermore, the role of income (especially that of women's poverty) has been hypothesized as a significant factor in the spread of HIV in SSA, but again there is no credible evidence showing a causal link between income and HIV risk. A randomized intervention, such as the one proposed here, that provides randomly varied amounts of cash transfers to young individuals and their guardians is the perfect setting to examine the possible existence of such causal relationships.

Objectives:

The objective of the proposed study here is to provide credible evidence on issues about which we still know very little. Specifically, the main questions the study will try to answer are the following:

1. Are the observed effects of a CCT associated with the transfer or the conditionality imposed on the recipient?
2. Do the outcomes of interest improve with increased benefit levels set by the program?
3. Do CCT programs for schooling have any positive health impacts, including prevention of STIs such as HIV/AIDS among young people?

ELIGIBILITY:
Inclusion Criteria:

* female
* 13-22 years old
* never married

Ages: 13 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3796 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Sexually Transmitted Infections | 18 months
  HIV prevalence HSV-2 prevalence
Schooling | 12 months/24 months
  school enrollment

SECONDARY OUTCOMES:
Sexually Transmitted Infections | 18 months
  syphilis
Marriage and fertility | 12 months/24 months
  ever married currently pregnant
sexual behavior | 12 months/ 24 months
  new sexual debut unprotected sexual intercourse weekly sexual intercourse had a sexual partner 25 or older
HIV Awareness | 12 months/24 months
  ever tested for HIV received health training on HIV HIV knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Berk Ozler, PhD, Principal Investigator — World Bank; Craig T McIntosh, PhD, Principal Investigator — University of California, San Diego; Sarah J Baird, PhD, Principal Investigator — George Washington University; Ephraim Chirwa, PhD, Principal Investigator — University of Malawi; Richard S Garfein, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Zomba District, Malawi, Zomba, Malawi

REFERENCES:
- [Result] Baird S, Chirwa E, McIntosh C, Ozler B. The short-term impacts of a schooling conditional cash transfer program on the sexual behavior of young women. Health Econ. 2010 Sep;19 Suppl:55-68. doi: 10.1002/hec.1569. PMID 19946887
- [Derived] Baird SJ, Garfein RS, McIntosh CT, Ozler B. Effect of a cash transfer programme for schooling on prevalence of HIV and herpes simplex type 2 in Malawi: a cluster randomised trial. Lancet. 2012 Apr 7;379(9823):1320-9. doi: 10.1016/S0140-6736(11)61709-1. Epub 2012 Feb 15. PMID 22341825